CLINICAL TRIAL: NCT00005272
Title: Smoking and Body Weight: Analysis of HHANES
Status: Completed | Type: Observational
Sponsor: University of Memphis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1157; R03HL046117 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To evaluate the relationships between smoking rate, gender, and body weight in the Hispanic Health and Nutrition Examination I Survey (HHANES) I. Also, to evaluate the independent and additive contribution of smoking rate and fasting glucose on body weight in HHANES I and NHANES II.

DETAILED DESCRIPTION:
BACKGROUND:

The study was supported by the Small Grants Program established by the National Heart, Lung, and Blood Institute in January 1990 to provide limited support to extend analyses of research data generated by clinical trials, population research, and demonstration and education research studies.

DESIGN NARRATIVE:

The first study used HHANES I data and analysis of variance to determine the possible body composition differences between subgroups of gender and smoking categories. Caloric differences in dietary intake were analyzed in a second ANOVA design.

The second study used data from HHANES I and NHANES II to evaluate the independent and additive or synergistic contribution of smoking rate and fasting glucose on body weight.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-09; Study Completion 1992-09

REFERENCES:
- [Background] Klesges RC, Klesges LM, Meyers AW. Relationship of smoking status, energy balance, and body weight: analysis of the Second National Health and Nutrition Examination Survey. J Consult Clin Psychol. 1991 Dec;59(6):899-905. doi: 10.1037//0022-006x.59.6.899. PMID 1774374
- [Background] Klesges RC, Ray JW, Klesges LM. Caffeinated coffee and tea intake and its relationship to cigarette smoking: an analysis of the Second National Health and Nutrition Examination Survey (NHANES II). J Subst Abuse. 1994;6(4):407-18. doi: 10.1016/s0899-3289(94)90334-4. PMID 7780298
- [Background] Klesges RC, Klesges LM. The relationship between body mass and cigarette smoking using a biochemical index of smoking exposure. Int J Obes Relat Metab Disord. 1993 Oct;17(10):585-91. PMID 8242127
- [Background] Klesges RC, Debon M, Ray JW. Are self-reports of smoking rate biased? Evidence from the Second National Health and Nutrition Examination Survey. J Clin Epidemiol. 1995 Oct;48(10):1225-33. doi: 10.1016/0895-4356(95)00020-5. PMID 7561984